CLINICAL TRIAL: NCT07129473
Title: Hyperemesis Gravidarum Risk Reduction With Metformin
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: The Morning Sickness & HG Clinic (Unknown)
Responsible Party: Principal Investigator, Marlena Fejzo, Clinical Assistant Professor of Population and Public Health Sciences in the Center for Genetic Epidemiology, University of Southern California
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APP-25-03192
Record Dates: First submitted 2025-08-07; First posted 2025-08-19 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Hyperemesis Gravidarum
Keywords: Metformin; HG; Hyperemesis; Hyperemesis Gravidarum; Nausea and Vomiting of Pregnancy; NVP; severe Nausea and Vomiting of Pregnancy; sNVP; Nausea; Vomiting; Pregnancy; Pregnant; Morning Sickness
MeSH Terms: conditions — Hyperemesis Gravidarum; Nausea; Vomiting; Morning Sickness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm (Experimental): Treatment Arm (N=112):
  * Individuals with a prior HG pregnancy with intravenous (IV) fluid treatment and current pregnancy intent
  * Residing in California or Alabama
  * Daily metformin-XR, escalated from 500 mg to 2000 mg as tolerated
  * Continue treatment until either 2 weeks post-pregnancy confirmation or up to 12 months
  Interventions: Drug: Metformin Extended Release Oral Tablet
- Survey/Comparator Arm (No Intervention): Survey/Comparator Arm (N=112):
  * Matched controls (race/ethnicity, parity, maternal age, prior HG pregnancy (IV fluids), pregnancy intent)
  * No metformin treatment

INTERVENTIONS:
Drug: Metformin Extended Release Oral Tablet — Participants in the Treatment Arm will receive oral extended-release metformin (metformin-XR) 1x daily with an evening meal starting prior to conception. Daily dosing will begin at 500 mg and increase gradually over an 8 week period (+500mg every 2 weeks, as tolerated) to a maximum tolerated dose of up to 2,000 mg. Treatment at highest tolerated dose will continue until either 2 weeks after a positive pregnancy test or 12 months from treatment start, whichever comes first. Participants will attend 3 clinic visits and provide blood samples at baseline, after dose escalation, and during early pregnancy to assess biomarker levels and genetic characteristics. Daily dosing, adherence, and side effects are recorded via MyCap; clinical visits include vital signs, PUQE-24/HELP scores, and blood draws (CBC, creatinine, genotyping, biomarker levels). Postpartum surveys include a metformin treatment & HG outcomes survey (REDCap) and additional measures (PES, MAPP-QOL, EPDS, PSAS, and ASQ-3).
  Arms: Treatment Arm

SUMMARY:
The goal of this clinical trial is to evaluate whether daily oral metformin extended-release (metformin-XR), taken prior to pregnancy, can reduce the risk and severity of Hyperemesis Gravidarum (HG)-a severe nausea and vomiting condition in pregnancy-in individuals aged 18-49 who have experienced HG in a previous pregnancy and are trying to conceive. Researchers also aim to better understand which individuals may respond well-or poorly-to metformin based on biological and clinical characteristics.

The main questions this study aims to answer are:

1. Is metformin-XR acceptable and well-tolerated when taken by non-pregnant individuals who have had HG in a previous pregnancy and are currently trying to conceive?
2. How safe and tolerable is metformin-XR when taken at increasing doses over 8 weeks and continued through early pregnancy (or for up to 12 months if pregnancy does not occur)?
3. Among those who become pregnant during the study, does pre-pregnancy metformin-XR use reduce the risk of HG coming back and lower the severity of nausea and vomiting symptoms?
4. How does pre-pregnancy metformin-XR use affect pregnancy outcomes, postpartum health, and newborn health and development?
5. Are there specific genetic, biomarker, demographic, or clinical features that predict whether someone is likely to benefit from metformin-XR or experience side effects that lead them to stop taking it?

Researchers will compare a metformin treatment group to a survey-only group (comparator) to see if metformin-XR is associated with improved outcomes, including reduced HG recurrence and better maternal and neonatal health indicators.

Participants will:

Complete online questionnaires before pregnancy, during early pregnancy, and postpartum

(Treatment group only) Take daily metformin-XR and attend three brief study visits

(Treatment group only) Undergo blood draws at specified timepoints to assess safety and biological response

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-49
* HG in prior pregnancy (clinical criteria: intravenous (IV) fluid treatment)
* Trying to conceive
* Willing to participate in a trial that includes daily use of an oral agent prior to pregnancy
* Treatment Arm: residing in California/Alabama
* Treatment Arm: normal blood panel (CBC) (e.g., white count, hemoglobin, platelets all within the normal range)
* Treatment Arm: normal creatinine levels (GFR < 45)
* Survey/Comparator Arm: not currently taking metformin and do not plan to take metformin during study period
* Able and willing to provide written informed consent prior to initiation of any study procedures.
* Demonstrates understanding of the study objectives, requirements, potential risks, and willingness to comply with study procedures and follow-up.

Exclusion Criteria:

* Allergic or adverse reaction to metformin-XR
* Chronic diseases/conditions
* Daily medications/substances (tobacco, cyclobenzaprine, cannabis, escitalopram, sertraline, other Selective Serotonin Reuptake Inhibitors (SSRIs))
* Assisted Reproductive Technology
* Pregnant
* Not trying to conceive
* Pre-existing kidney dysfunction
* Treatment Arm: Residing outside California/Alabama
* Anemia
* Treatment Arm: abnormal blood panel (CBC) (e.g., white count, hemoglobin, or platelets not within the normal range)
* Treatment Arm: abnormal creatinine levels (GFR > 45 excluded from the study, signs of kidney disease)
* Survey/Comparator Arm: current metformin use or plans to take metformin during study period
* Not able and willing to provide written informed consent prior to initiation of any study procedures.
* Does not demonstrate understanding of the study objectives, requirements, potential risks, and willingness to comply with study procedures and follow-up.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 224 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2030-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Adherence to Escalating Doses of Metformin-XR | Baseline to 8 weeks after treatment initiation
  Proportion of participants in the Treatment Arm who reach and maintain each target dose level during the 8-week dose-escalation period, as recorded via MyCap survey entries.
Tolerability and Safety of Metformin-XR | Baseline through treatment completion (up to 12 months after treatment initiation or 2 weeks after confirmed pregnancy, whichever comes first)
  Number and severity of treatment-related adverse events and dose-limiting toxicities experienced by participants during the 8-week dose-escalation period and maintenance phase. Safety assessed by participant report, clinical evaluations, and laboratory results.
Hyperemesis Gravidarum (HG) Recurrence and Severity | From confirmed pregnancy through 12 weeks of gestation
  Incidence and severity of HG in subsequent pregnancy, assessed using validated tools (Pregnancy-Unique Quantification of Emesis (PUQE-24), HyperEmesis Level Prediction (HELP) Score) and pregnancy experience survey responses.
Pregnancy & Neonatal Outcomes: Incidence of Pregnancy Complications | From confirmed pregnancy through delivery
  Proportion of participants who experience predefined pregnancy complications (e.g., gestational diabetes, preeclampsia, gestational hypertension). Data will be abstracted from medical records and study surveys.
Pregnancy & Neonatal Outcomes: Delivery Characteristics | At delivery
  Proportion of participants with a favorable delivery outcome, defined as live birth at ≥37 weeks gestation. Delivery outcome will be abstracted from medical records and study surveys.
Pregnancy & Neonatal Outcomes: Assessment of Peripartum Events | From confirmed pregnancy to 6 months postpartum
  Peripartum events will be evaluated using the validated Peripartum Events Scale (PES). PES score will be evaluated via medical record abstraction. The lowest possible PES score is zero, with higher scores corresponding to more stressful labor and delivery experiences.
Pregnancy & Neonatal Outcomes: Maternal Postpartum Depression | From birth to 6 months postpartum
  Maternal mental health will be assessed using the Edinburgh Postnatal Depression Scale (EPDS). The EPDS range is 0-30, with higher scores corresponding to more severe depressive symptoms.
Pregnancy & Neonatal Outcomes: Maternal Postpartum Anxiety | From birth to 6 months postpartum
  Maternal mental health will be assessed using the Postpartum-Specific Anxiety Scale (PSAS). The PSAS range is 51-204, with higher scores corresponding to greater postpartum-specific anxiety.
Pregnancy & Neonatal Outcomes: Maternal Postpartum Quality of Life | From birth to 6 months postpartum
  Maternal postpartum quality of life will be assessed using the validated Maternal Postpartum Quality of Life (MAPP-QOL) Questionnaire. The MAPP-QOL possible total score range is 38-228, with higher scores corresponding to better quality of life.
Pregnancy & Neonatal Outcomes: Neonatal Health Status | At delivery
  Proportion of neonates who experience an adverse neonatal outcome, defined as the presence of at least one predefined adverse neonatal event, including but not limited to low birth weight (<2500 grams), preterm birth (<37 weeks gestation), admission to a neonatal intensive care unit (NICU), or low 5-minute Apgar score (<7). Data will be obtained from medical record abstraction and study surveys.
Pregnancy & Neonatal Outcomes: Child Developmental Status | From birth to 6 months postpartum (with optional follow up until the end of the 5-year study period)
  Child development will be assessed before 6 months postpartum using the validated Ages and Stages Questionnaires, Third Edition (ASQ-3). Optionally, every 6 months up to year 5 (study completion), participants will have the opportunity to complete an additional ASQ-3 assessment corresponding to their child's age to report long-term child outcomes.
Indicators of Metformin Response: Genetic Factors | Once at baseline
  Genotyping of variants associated with HG risk (e.g., rs1058587/GDF15, rs9312688/IGFBP7, rs12790159/PGR, and rs10948901/GFRAL) to explore their association with metformin response and pregnancy outcomes.
Indicators of Metformin Response: Circulating Biomarker Levels | Once at baseline, once when participant reaches highest tolerated metformin dose (up to week 8), and once at pregnancy confirmation in participants who conceive
  Measurement of biomarker (e.g., GDF15, IGFBP7) concentrations at three timepoints in the Treatment Arm (baseline, after dose escalation, and during early pregnancy) to explore the role of each as a predictive biomarker for HG and metformin response.
Indicators of Metformin Response: Demographic Characteristics | At baseline
  Demographic information will be collected via initial study survey and qualitatively analyzed for associations with HG and metformin response.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fejzo M, Rocha N, Cimino I, Lockhart SM, Petry CJ, Kay RG, Burling K, Barker P, George AL, Yasara N, Premawardhena A, Gong S, Cook E, Rimmington D, Rainbow K, Withers DJ, Cortessis V, Mullin PM, MacGibbon KW, Jin E, Kam A, Campbell A, Polasek O, Tzoneva G, Gribble FM, Yeo GSH, Lam BYH, Saudek V, Hughes IA, Ong KK, Perry JRB, Sutton Cole A, Baumgarten M, Welsh P, Sattar N, Smith GCS, Charnock-Jones DS, Coll AP, Meek CL, Mettananda S, Hayward C, Mancuso N, O'Rahilly S. GDF15 linked to maternal risk of nausea and vomiting during pregnancy. Nature. 2024 Jan;625(7996):760-767. doi: 10.1038/s41586-023-06921-9. Epub 2023 Dec 13. PMID 38092039
- [Background] Sharma N, MacGibbon KW, Brecht-Doscher A, Cortessis VK, Fejzo MS. Prepregnancy metformin use associated with lower risk of severe nausea and vomiting of pregnancy and hyperemesis gravidarum. Am J Obstet Gynecol. 2025 Dec;233(6):649.e1-649.e14. doi: 10.1016/j.ajog.2025.06.055. Epub 2025 Jun 28. PMID 40588059